CLINICAL TRIAL: NCT01268007
Title: This is an Observational, Un-blinded, Non-significant Risk, Non-interventional Study Designed to Collect ECG Data on at Least One Subject Out of a Pool of up to Three (3) Healthy Male Subjects at One Clinical Site (Clinical Trials of Texas).
Brief Title: Heartbeat Sensitivity Calibration Using the ECG Accessory
Status: Completed | Type: Observational
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Dr. Douglas Denham, DO, Clinical Trials of Texas
Other Study IDs: E-46
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2010-12

CONDITIONS: ECG Comparisons in Normal Healthy Subject

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Normal ECG measurements: Observational, un-blinded, non-interventional study designed to collect ECG data on at least one (1) male patient in an outpatient setting.

SUMMARY:
This is an observational, un-blinded, non-significant risk, non-interventional study designed to collect ECG data on at least one subject out of a pool of up to three (3) healthy male subjects at one clinical site (Clinical Trials of Texas). Cyberonics will be collecting ECG recordings collected by an investigational device for comparison with conventional ECG recordings. This data will be used to validate a new device under development.

DETAILED DESCRIPTION:
This is an observational, un-blinded, non-significant risk, non-interventional study designed to collect ECG data on at least one subject out of a pool of up to three (3) healthy male subjects at one clinical site (Clinical Trials of Texas). If acceptable data is acquired from one (1) subject the remaining subjects will not be entered into the study. Three (3) to six (6) researchers will record data, but all direct contact with the subject will be done by the study coordinator or principal investigator (PI).

The purpose of this study is to validate a Heartbeat Sensitivity calibration process utilizing the Cyberonics ECG Accessory. The non-invasive, passive collection of ECG signals from a resting healthy subject will be used to validate the use of the ECG Accessory with the Model 201 Programming Wand, Model 250 VNS Programming Software Version 9.0, Model 106 Generator, and ECG monitor (DRE True ECG-12), as well as the associated Instructions for Use. The data generated from this exercise will be used in future clinical trials utilizing this device.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients must be 18 years or older, male, and of any race.
* 2. Patient must be in good general health, fully ambulatory, and able to complete the physical aspects of testing requirements.
* 3. Patient must be willing and able to complete informed consent and HIPAA authorization.

Exclusion Criteria:

* 1. Subjects with skin abnormalities or conditions that would interfere with ECG electrode patch placement or cause subject discomfort with patch placement.
* 2. Subjects report history of allergies or sensitivity to adhesive tapes or patches.
* 3. Subjects with major health condition that in the investigator's judgment would prevent the subject's successful completion of the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal Healthy male
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2010-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Comparison of ECG measurements | 8 hours
  No specific effectiveness outcomes or calculations are planned for this non-interventional study. The sponsor will use the ECG data collected during this study as a comparison of the subject's actual ECG waveforms obtained through standard ECG connections to the ECG Accessory transmitted heart beat detection signals from the Model 106 Generator to the ECG monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials of Texas, San Antonio, Texas, United States